CLINICAL TRIAL: NCT02564666
Title: The Effect of Telephone Counseling on the Compliance and the Level of Satisfaction for Patients Receiving Sorafenib Due to Advanced Hepatocellular Carcinoma
Brief Title: The Effect of Telephone Counseling on the Compliance and Satisfaction for Advanced HCC Patients Receiving Sorafenib
Acronym: SORATEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ju Hyun Shim, Prof., Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2015-0815
Record Dates: First submitted 2015-08-20; First posted 2015-10-01 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; sorafenib; telephone counseling
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telephone counseling (Active Comparator): regular telephone counseling per week
  Interventions: Other: telephone counseling
- No telephone counseling (No Intervention): no regular telephone counseling

INTERVENTIONS:
Other: telephone counseling — regular telephone counseling for compliance and advese event
  Arms: Telephone counseling

SUMMARY:
Sorafenib is an oral multikinase inhibitor with antiproliferative and antiangiogenic effects used as systemic treatment in patients with unresectable hepatocellular carcinoma.

Although sorafenib has demonstrated many clinical benefits in patients, its adverse cannot be ignores.

This drug occasionally causes severe adverse events (AEs), which include hand-foot skin reaction (HFSR), hypertension, diarrhea, anorexia, fatigue, weight loss, and so on. Although most adverse events are reversible, they can significantly impact a patient's quality of life and occasionally result in dose reduction or discontinuation of therapy Patients are also more likely to remain on treatment if they are guided over the difficult initial 4~6wks of therapy during which time the development of adverse events following sorafenib treatment initiation are most likely to occur.

Patient education, proactive management and establishing and maintaining open communication between patients and the nurse are crucial to the effective management of these adverse events.

This study design is a randomized controlled trial and 64 patients will be randomized to one of 2 groups in a 1:1 ratio. 32 patients will be enrolled into the controlled group and the rest of 32 patients will be enrolled into the intervention group. The intervention group will be received the routine telephone calls of six times at intervals of once a week during 10~15 minutes (from a well-trained nurse)

The purpose of this study is to confirm whether an effective intervention that telephone counseling and education by a nurse can increase drug compliance for patients with HCC who is taking Sorafenib and is to use for developing individual educational program as a fundamental data that can be applied for patients taking Sorafenib after investigating patient satisfaction by "The Satisfaction with information about Medicines Scale(SIMS)" tool.

DETAILED DESCRIPTION:
This study design is a randomized controlled trial and 64 patients will be randomized to one of 2 groups in a 1:1 ratio. 32 patients will be enrolled into the controlled group and the rest of 32 patients will be enrolled into the intervention group. The intervention group will be received the routine telephone calls of six times at intervals of once a week during 10~15 minutes (from a well-trained nurse)

The purpose of this study is to confirm whether an effective intervention that telephone counseling and education by a nurse can increase drug compliance for patients with HCC who is taking Sorafenib and is to use for developing individual educational program as a fundamental data that can be applied for patients taking Sorafenib after investigating patient satisfaction by "The Satisfaction with information about Medicines Scale(SIMS)" tool.

ELIGIBILITY:
Inclusion Criteria:

* Patient who agrees voluntarily
* Patient with a diagnosis of HCC is receiving Sorafenib monotherapy.
* Child-Pugh class, A or B, ECOG PS 0~2
* 20 years of age or older.
* Patient who can listen and speak Korean

Exclusion Criteria:

* lack of cognitive ability or any r psychiatric illness
* Patient who is receiving combination treatment of TACE or other HCC treatment with Sorafenib.
* A hearing-impaired patient.
* Patient who has accompanied other primary malignants tumor in other organs except for HCC.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Drug compliance for patients with HCC who is taking Sorafenib compliance | 6 weeks
  "Drug compliance for patients with HCC who is taking Sorafenib" as Assessed by MMAS-8 Score and compare "MMAS-8 score" between control group and intervention group.
  Measurement is Scores range from 0 [high adherence] to 3~8 [low adherence] )

SECONDARY OUTCOMES:
Survival rate | 12 months
Duration of dosing period | 12 months

OTHER OUTCOMES:
The satisfaction with Information about Medicines Scale (SIMS) score | 6 weeks
  SIMS is to use for developing individual educational program as a fundamental data that can be applied for patients taking Sorafenib

CONTACTS AND LOCATIONS:
Overall Officials: Ju Hyun Shim, MD. PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea